CLINICAL TRIAL: NCT03734991
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral Ibrexafungerp (SCY-078) vs. Placebo in Subjects With Acute Vulvovaginal Candidiasis
Brief Title: Efficacy and Safety of Oral Ibrexafungerp (SCY-078) vs. Placebo in Subjects With Acute Vulvovaginal Candidiasis (VANISH 303)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCY-078-303
Record Dates: First submitted 2018-10-30; First posted 2018-11-08 (Actual); Results first posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Candida Vulvovaginitis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: randomized, placebo-controlled, double-blind study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ibrexafungerp (SCY-078) (Experimental): 300 mg orally every 12 hrs for 1 day (2 doses in 1 day)
  Interventions: Drug: Ibrexafungerp
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibrexafungerp — Ibrexafungerp 300 mg BID for 1 day
  Other Names: SCY-078
  Arms: Ibrexafungerp (SCY-078)
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, multicenter, double-blind, placebo-controlled study to evaluate the efficacy and safety of oral Ibrexafungerp (SCY-078) compared to placebo in female subjects 12 years and older with AVVC.

DETAILED DESCRIPTION:
Subjects who meet all of the inclusion and none of the exclusion criteria will be enrolled into the study and will be randomized in a 2:1 ratio to either oral ibrexafungerp or ibrexafungerp matching placebo, as follows:

* Oral ibrexafungerp 300-mg dose BID for 1 day
* Oral ibrexafungerp matching placebo BID for 1 day

Subjects will receive their first dose of study drug at the site and will be dispensed the second dose for self-administration at home 12 hours after the first dose. Study Blinding, Randomization and Stratification: This is a randomized, double-blind study.

All site and sponsor personnel will be blinded to treatment assignment. Approximately 366 eligible subjects will be enrolled and randomized in a 2:1 ratio to one of the two study treatment groups. For the purpose of maintaining treatment blinding, all subjects randomized to the placebo group will receive matching ibrexafungerp placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

Subject is a postmenarchal female subject 12 years and older

Subject has a diagnosis of symptomatic AVVC at baseline including a positive microscopic examination with 10% KOH in a vaginal sample revealing yeast forms (hyphae/pseudohyphae) or budding yeasts, and vaginal pH (≤4.5)

Exclusion Criteria:

Subject has any vaginal condition other than AVVC that may interfere with the diagnosis or evaluation of response to therapy, such as suspected or confirmed concurrent causes of vulvovaginitis and/or cervicitis (mixed infection)

Need for systemic and/or topical (vaginal) antifungal treatment, including prescription or over-the-counter products during the study and treatment for VVC 28 days prior to randomization

Subject is actively menstruating at the time of the Baseline visit.

Subject has uncontrolled diabetes mellitus.

Subject has a vaginal sample with pH >4.5.

Subject has a history of or an active cervical/vaginal cancer.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 376 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Womens' Health Care Research Corp, San Diego, California
  - Women's Medical Research Group, Clearwater, Florida
  - Altus Research, Lake Worth, Florida
  - OBGYN Assoc of Mid Florida, Leesburg, Florida
  - New Age Medical Research Corporation, Miami, Florida
  - Clinical Trials Management LLC, Covington, Louisiana
  - Clinical Trials Management LLC, Metairie, Louisiana
  - Unified Women's Clinical Research- Hagerstown, Hagerstown, Maryland
  - Wayne State University, Detroit, Michigan
  - Consultants In Women's Healthcare, Inc., St Louis, Missouri
  - Center For Women's Health and Wellness LLC - Interspond - PPDS, Lawrenceville, New Jersey
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - GYN Center for Women PA, Durham, North Carolina
  - Carolina Women's Research and Wellness Center, Durham, North Carolina
  - Unified Women's Clinical Research Greensboro, Greensboro, North Carolina
  - Unified Women's Clinical Research, Morehead City, North Carolina
  - Unified Women's Clinical Research Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research - Lyndhurst Clinical Research, Winston-Salem, North Carolina
  - Medical Research South, Charleston, South Carolina
  - Magnolia Ob/Gyn Research Center, LLC, Myrtle Beach, South Carolina
  - Medical Research Center of Memphis, Memphis, Tennessee
  - TMC Life Research Inc, Houston, Texas
  - Group For Women, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goje O, Sobel R, Nyirjesy P, Goldstein SR, Spitzer M, Faught B, Larson S, King T, Azie NE, Angulo D, Sobel JD. Oral Ibrexafungerp for Vulvovaginal Candidiasis Treatment: An Analysis of VANISH 303 and VANISH 306. J Womens Health (Larchmt). 2023 Feb;32(2):178-186. doi: 10.1089/jwh.2022.0132. Epub 2022 Oct 17. PMID 36255448

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral at 28 medical centers between 04Jan2019 and 04Sep2019.
Period: Overall Study
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Started | 249 | 127
Withdrawn Before Treatment | 2 | 3
Withdrawn Before TOC | 59 | 41
Completed the TOC Visit | 188 | 83
Withdrawn At or After the TOC Visit | 5 | 3
Completed | 183 | 80
Not Completed | 66 | 47
Not completed — Adverse Event | 4 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lack of efficacy and or/use of antifungal therapy | 49 | 41
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibrexafungerp (SCY-078) | Placebo | Total
Number analyzed (Participants) | 247 | 124 | 371
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 244 | 120 | 364
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.22) | 35.8 (12.47) | 34.9 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 124 | 371
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 25 | 89
  Not Hispanic or Latino | 183 | 99 | 282
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 101 | 51 | 152
  White | 132 | 71 | 203
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 247 | 124 | 371

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure (Complete Resolution of Signs and Symptoms)
Description: measured by the percentage of subjects with clinical cure (complete resolution of signs and symptoms) at the test-of-cure (TOC) visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 188 | 98
Participants
  Clinical cure | 95 | 28
  Clinical failure | 93 | 70

2. Secondary Outcome: Mycological Eradication (Negative Culture for Growth of Yeast)
Description: percentage of subjects with mycological eradication (negative culture for growth of Candida species) at the TOC visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 188 | 98
Participants
  Mycological eradication | 93 | 19
  Mycological persistence | 95 | 79

3. Secondary Outcome: Clinical Cure and Mycological Eradication (Responder Outcome)
Description: percentage of subjects with clinical cure and mycological eradication (responder outcome) at the TOC visit
Time Frame: Day 8-14
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 178 | 95
Participants
  Overall success | 64 | 12
  Overall failure | 114 | 83

4. Secondary Outcome: Complete Clinical Response at Follow-Up
Description: percentage of subjects with complete resolution of signs and symptoms at the Follow-up (FU) visit
Time Frame: Day 25
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 190 | 100
Participants
  Clinical cure at Follow up | 113 | 44
  Clinical failure at Follow up | 77 | 56

5. Secondary Outcome: Overall Treatment-Emergent Adverse Events (Safety Set)
Description: Number of subjects with treatment related adverse events
Time Frame: Up to 29 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
Number analyzed (Participants) | 247 | 124
Participants
  Any treatment-emergent, treatment-related adverse event | 98 | 21
  No treatment-emergent, treatment-related adverse events | 149 | 103

ADVERSE EVENTS:
Time Frame: 4 weeks after last dose
Arm/Group | Ibrexafungerp (SCY-078) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/124
Serious Adverse Events (participants affected / at risk) | 1/247 | 2/124
Other Adverse Events (participants affected / at risk) | 117/247 | 34/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (SCY-078) (N=247) | Placebo (N=124)
Hypokalaemia (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Pneumonia and bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp (SCY-078) (N=247) | Placebo (N=124)
Diarrhoea (Gastrointestinal disorders) | 63 | 8
Nausea (Gastrointestinal disorders) | 40 | 7
Abdominal pain (Gastrointestinal disorders) | 17 | 3
Abdominal discomfort (Gastrointestinal disorders) | 14 | 2
Bacterial vaginosis (Infections and infestations) | 13 | 10
Headache (Nervous system disorders) | 23 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT03734991/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03734991/SAP_001.pdf